CLINICAL TRIAL: NCT00234052
Title: Phase II Trial of Carboplatin and Pemetrexed Plus Bevacizumab in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Carboplatin, Pemetrexed Disodium, and Bevacizumab in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04L2; NU-04L2; STU00007415 (Other: Northwestern University IRB#)
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Carboplatin; Pemetrexed

ARMS (1):
- Treatment Arm (Experimental): Carboplatin + pemetrexed + bevacizumab
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: pemetrexed

INTERVENTIONS:
Biological: bevacizumab — 5 mg/kg administered intravenously over 90 minutes on day 1 of each cycle (cycle = 3 weeks)
  Other Names: Avastin
Drug: carboplatin — Administered intravenously at a dose of AUC=6 over 30 minutes on day 1 of each cycle (1 cycle = 3 weeks)
Drug: pemetrexed — Administered intravenously at a dose of 500 mg/m2 over 10 minutes on day 1 of each cycle (1 cycle = 3 weeks)
  Other Names: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving carboplatin and pemetrexed disodium together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin and pemetrexed disodium together with bevacizumab works in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the median time to disease progression in patients with stage IIIB or IV or recurrent non-squamous cell non-small cell lung cancer treated with carboplatin, pemetrexed disodium, and bevacizumab.

Secondary

* Determine the response rate and duration of response in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients with complete response, partial response, or stable disease continue to receive pemetrexed disodium and bevacizumab in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or cytologically* confirmed non-small cell lung cancer

  * Any histology, except squamous cell carcinoma, allowed

    * Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible
  * No histology in close proximity to a major vessel or cavitation NOTE: *Histologic or cytologic elements may be established on metastatic tumor aspirates or biopsy
* Meets 1 of the following stage criteria:

  * Stage IIIB disease (with malignant pleural effusion)
  * Stage IV disease
  * Recurrent disease
* Measurable or non-measurable disease
* No known CNS metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* No history of hemorrhagic disorders

Hepatic

* Bilirubin < 1.5 mg/dL
* AST and ALT < 5 times upper limit of normal
* INR < 1.5
* PTT normal

Renal

* Creatinine clearance ≥ 45 mL/min
* Urine protein:creatinine ≤ 1.0 by spot urinalysis

Cardiovascular

* No myocardial infarction within the past 6 months
* No New York Heart Association class II-IV congestive heart failure
* No unstable angina pectoris
* No serious cardiac arrhythmia requiring medication
* No stroke within the past 6 months
* No peripheral vascular disease ≥ grade 2
* No uncontrolled hypertension (i.e., blood pressure ≥ 150/100 mm Hg)

  * Patients with a history of hypertension allowed provided blood pressure is well controlled on a stable regimen of anti-hypertensive therapy
* No history of thrombotic disorders
* No other clinically significant cardiovascular disease

Pulmonary

* No history of gross hemoptysis, defined as bright red blood of a ½ teaspoon or more

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be willing and able to take daily oral folic acid, intermittent vitamin B_12 injections, and corticosteroid premedication
* No ongoing or active infection
* No serious, non-healing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 3 weeks since prior immunotherapy

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* More than 3 weeks since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* More than 3 weeks since prior radiotherapy

Surgery

* More than 4 weeks since prior major surgery
* More than 1 week since prior minor surgery, fine needle aspiration, or core biopsy
* No concurrent major surgery

Other

* Recovered from all prior therapy
* More than 4 weeks since prior and no concurrent participation in another experimental drug study
* No aspirin or other nonsteroidal anti-inflammatory drug (NSAID) 2 days before and 2 days after each pemetrexed disodium infusion (5 days before and 2 days after each pemetrexed disodium infusion for NSAIDs with a long half-life [e.g., naproxen, rofecoxib, or celecoxib])
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic anticoagulation for venous access devices allowed provided requirements for INR and PTT are met
* No concurrent administration of any of the following:

  * Chronic daily treatment with aspirin (> 325 mg per day)
  * NSAIDs known to inhibit platelet function, including any of the following:

    * Dipyridamole
    * Ticlopidine
    * Clopidogrel
    * Cilostazol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-07-28 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti D. Patel, Study Chair — Robert H. Lurie Cancer Center
Locations (5):
- United States (5):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on June 1, 2005 with an accrual goal of 50 patients. The first patient enrolled started treatment on July 28, 2005. The study was closed permanently on July 10, 2007 when accrual had been met with 51 patients registered and 50 patients treated on study.
Groups:
- Treatment With Carboplatin + Pemetrexed + Bevacizumab: Carboplatin + Pemetrexed + Bevacizumab
  Patients will receive 6 cycles where (1 cycle is 21 days) of :
  Bevacizumab: 15 mg/kg administered intravenously over 30 - 90 minutes on day 1 of each cycle Carboplatin: Administered intravenously at a dose of AUC=6 over 30 minutes on day 1 of each cycle Pemetrexed: Administered intravenously at a dose of 500 mg/m2 over 10 minutes on day 1 of each cycle
  Patients without progression will go into the maintenance phase and receive cycles of the following where 1 cycle is 21 days:
  Bevacizumab: 15 mg/kg administered intravenously over 30 - 90 minutes on day 1 of each cycle Pemetrexed: Administered intravenously at a dose of 500 mg/m2 over 10 minutes on day 1 of each cycle
Period: Treatment
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Started | 51
Started Treatment | 50
Completed 6 Cycles | 33
Went Into Maintenance Phase | 30
Completed | 30
Not Completed | 21
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 5
Not completed — Death | 2
Not completed — Progressive Disease | 11
Period: Follow-up for 5 Years
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Started | 50 (All patients that are treated on study go into the follow up period.)
Completed | 1
Not Completed | 49
Not completed — Death | 41
Not completed — Lost to Follow-up | 1
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 41
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival
Description: Progression Free Survival (PFS) in patients treated with the combination of carboplatin, pemetrexed and bevacizumab is defined as the time from registration to the time of documented disease progression or death from any cause. Patients that were lost to follow up or withdrew consent were censored at that point.
Time Frame: Approximately every 3 weeks until disease progression or death. Median follow up of 13 months (range 0.8 to 34.4 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 50
Months | 7.8 [5.2 to 11.5]

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) of patients treated with carboplatin, pemetrexed, and bevacizumab combination is defined as the number of patients who's best response is a Complete Response (CR) plus Partial Response (PR)as recorded from the start of treatment until disease progression as assessed by RECIST 1.0.
  CR=Disappearance of all target lesions for a minimum of 4 weeks. PR=At least a 30% decrease in the sum of the longest diameter (LD) of target lesions for a minimum of 4 weeks, taking as reference the baseline sum LD. No simultaneous increase in the size of any lesion or the appearance of a new lesion may occur.
Time Frame: Every two cycles until disease progression. Median follow up of 13 months (range 0.8 to 34.4 months)
Population: One patient received less than one cycle and was determined to not be evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 49
Participants | 27

3. Secondary Outcome: Toxicity of Carboplatin, Pemetrexed and Bevacizumab Combination Treatment
Description: To characterize the toxicity profile of carboplatin, pemetrexed and bevacizumab combination treatment.
  Toxicity data will be collected from initiation of treatment, every cycle, until 30 days post last treatment. Adverse events will be graded according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). Only toxicity determined to be a least possibility related to at least one study drug and grade 3 or 4 was collected for this outcome measure.
  In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: From treatment initiation, at the beginning of each cycle where one cycle equals 21 days until 30 days post treatment (range of cycles 1-51)
Population: This includes AEs observed before there was an amendment of the protocol to exclude patients with histories of diverticulitis or clinically significant diverticular disease. Any patient that received one dose of study drug is evaluable for this objective.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 50
Participants
  Anemia | 3
  Thrombocytopenia | 4
  Neutropenia | 2
  Venous Thrombosis | 3
  Fatigue | 4
  Diverticulitis | 4
  Infection | 5
  Proteinuria | 1
  Arterial Thrombosis | 1
  Increased Creatinine Levels | 1

4. Secondary Outcome: Overall Survival Rate
Description: Overall Survival (OS) Rate of carboplatin, pemetrexed and bevacizumab combination treatment is defined from the time of registration to the study until death from any cause. Patients that are lost to follow up will be censored from last documentation of survival status.
Time Frame: During treatment and then every 3 months x 2 years, then every 6 months x 3 years or until death.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 50
Months | 14.1 [10.6 to 19.6]

5. Secondary Outcome: Duration of Response
Description: Duration of Response for patients treated with the combination of carboplatin, pemetrexed and bevacizumab is measured from the time measurement criteria are met for Complete Response or Partial Response (whichever is first recorded) until the first date of documented progressive disease.
Time Frame: From documentation of response, every two cycles (1 cycle = 21 days) until progressive disease with range of cycles completed 1-51.
Population: Patients with response were included in this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 27
Months | 7.7 [4.4 to 12.5]

6. Post Hoc Outcome: Progression Free Survival at 6, 12, 18, 24 Months
Description: Progression Free Survival (PFS) Rate of carboplatin, pemetrexed and bevacizumab combination treatment is defined as the percentage of patients without progression at the following time points from registration to the study:
  6 months 12 months 18 months 24 months.
Time Frame: 6, 12,18, and 24 months from treatment initiation
Population: One patient received less than one cycle and was determined to not be evaluable for this objective.
Measure: Number; unit: percentage of patients with PFS
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 50
percentage of patients with PFS
  6 Months | 59
  12 Months | 34
  18 Months | 27
  24 Months | 19

7. Post Hoc Outcome: Overall Survival Rate at 6, 12, 18, and 24 Months
Description: Overall Survival (OS) Rate of carboplatin, pemetrexed and bevacizumab combination treatment will be defined as the percentage of patients with documentation of status of alive at the following timepoints from registration to the study:
  6 months 12 months 18 months 24 months
Time Frame: 6, 12,18, and 24 months from treatment initiation
Measure: Number; unit: percentage of patients alive
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
Number analyzed (Participants) | 50
percentage of patients alive
  6 Months | 86
  12 Months | 61
  18 Months | 38
  24 Months | 26

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment, every cycle, until 30 days post the last treatment where one cycle equals 21 days. Range of cycles completed by patients = 1 cycle to 51 cycles.
Arm/Group | Treatment With Carboplatin + Pemetrexed + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 41/50
Serious Adverse Events (participants affected / at risk) | 22/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Carboplatin + Pemetrexed + Bevacizumab (N=50)
Puesdogout (Musculoskeletal and connective tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Heart Attack (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Bowel Obstruction (Gastrointestinal disorders) | 1
Acute and Chronic Cholelithiasis (Gastrointestinal disorders) | 2
Diverticulitis (Gastrointestinal disorders) | 4 — Experienced before protocol amended to exclude patients with a history of diverticulitis
Vomiting (Gastrointestinal disorders) | 1 — Patient also with Nausea, Constipation and anemia
Epistaxis (General disorders) | 2
Osteomylitis of the right great toe (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Axillary Abscess (Infections and infestations) | 1
Seizures (Nervous system disorders) | 1
Viral Pneumonitis resulting in Death (Infections and infestations) | 1
Pneumonia/death (Infections and infestations) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Carboplatin + Pemetrexed + Bevacizumab (N=50)
Neutrophils (Neutropenia) (Blood and lymphatic system disorders) | 6
Hemoglobin (Anemia) (Blood and lymphatic system disorders) | 30
Leukocytes (Total white blood cells) (Blood and lymphatic system disorders) | 9
Platelets (Thrombocytopenia) (Blood and lymphatic system disorders) | 11
Hypertension (Cardiac disorders) | 20
Fatigue (General disorders) | 43
Fever (General disorders) | 4
Insomnia (General disorders) | 3
Weight Loss (General disorders) | 10
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6
Anorexia (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 12
Mucositis/Stomatitis (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 11
Epistaxis (Nosebleed) (General disorders) | 8
Urinary Tract Infection NOS (Renal and urinary disorders) | 3
Infection NOS (Infections and infestations) | 4
Alkaline Phosphastase Increase (Metabolism and nutrition disorders) | 8
Transaminase (Metabolism and nutrition disorders) | 6
ALT Increase (Metabolism and nutrition disorders) | 4
AST Increase (Metabolism and nutrition disorders) | 5
Albumin Decrease (Metabolism and nutrition disorders) | 5
Creatinine, Serum-high (Metabolism and nutrition disorders) | 9
Calcium, Serum-low (Hypocalcemia) (Metabolism and nutrition disorders) | 3
Glucose, Serum-high (Hyperglycemia) (Metabolism and nutrition disorders) | 18
Proteinuria (Metabolism and nutrition disorders) | 4
Neuropathy: Sensory (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Mood Alteration - Anxiety (Nervous system disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 9
Pain NOS (General disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Shortness of Breath) (Respiratory, thoracic and mediastinal disorders) | 24
Watery Eye (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No